CLINICAL TRIAL: NCT03447132
Title: Multicentre, International Neoadjuvant Randomized Double-blind Trial Comparing Fulvestrant® to a Combination of Fulvestrant® and Palbociclib (CDK 4/6 Inhibitor) in Patients With Operable Luminal Breast Cancer Responding to Fulvestrant®
Brief Title: Fulvestrant Versus Fulvestrant Plus Palbociclib in Operable Breast Cancer Responding to Fulvestrant
Acronym: SAFIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Cancer Research Group, United Arab Emirates (Other)
Collaborators: AstraZeneca (Industry); Pfizer (Industry); Genomic Health®, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICRG1201
Record Dates: First submitted 2018-02-11; First posted 2018-02-27 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2018-11

CONDITIONS: Breast Neoplasm Female
Keywords: Breast Cancer; Luminal; Neoadjuvant; pCR; Surgery
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; palbociclib; Goserelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fulvestrant 500mg + Palbociclib 125mg (Active Comparator): + Goserelin 3.6 mg if pre or peri menopausal patient - duration 4 months
  Interventions: Drug: Fulvestrant 500mg; Drug: Palbociclib 125mg; Drug: Goserelin 3.6 MG
- Fulvestrant 500mg + Placebos (Placebo Comparator): + Goserelin 3.6 mg if pre or peri menopausal patient - duration 4 months
  Interventions: Drug: Fulvestrant 500mg; Drug: Goserelin 3.6 MG; Drug: Placebos

INTERVENTIONS:
Drug: Fulvestrant 500mg — All patients in all arms will receive Fulvestrant 500mg
Drug: Palbociclib 125mg — Dose reduction to 100 mg and 75 mg
  Arms: Fulvestrant 500mg + Palbociclib 125mg
Drug: Goserelin 3.6 MG — Only for pre or peri menopausal patient
Drug: Placebos — Placebo
  Arms: Fulvestrant 500mg + Placebos

SUMMARY:
This is a multicenter, international, double-blind randomized Phase III study to evaluate the pathological complete response (pCR) according to Chevalier classification between Fulvestrant® and the combination of Fulvestrant® plus Palbociclib as neoadjuvant therapy of hormone-sensitive patients with operable luminal breast cancer.

Eligible patients will be assessed upfront using the OncotypeDX® molecular test (Recurrence Score <31).

DETAILED DESCRIPTION:
This is a multicenter, international, double-blind, randomized study.

Eligible patients based on inclusion/exclusion criteria will be assessed using OncotypeDX molecular test. Patients with low/intermediate risk (Recurrence Score <31) will be treated with the induction neoadjuvant Fulvestrant (500 mg (milligram) intra muscular(i.m) at Day 1, 14 and 28 and then every 4 weeks), plus Goserelin (3.6 mg subcutaneous (s.c) every 4 weeks, only for pre and peri-menopausal patients) for 4 months, followed by clinical and radiological assessment of the disease response.

Patients with objective response or stabilization will be randomized and treated for 4 additional months with:

* Fulvestrant 500 mg i.m every 4 weeks (+ Goserelin 3.6 mg s.c every 4 weeks, only for pre and peri-menopausal patients) and Placebo

or

* Combination Fulvestrant 500 mg i.m every 4 weeks (+ Goserelin 3.6 mg s.c every 4 weeks, only for pre and peri-menopausal patients) and Palbociclib 125 mg per os daily, 3 weeks on and 1 week off.

Patients with documented progressive disease will be considered at the discretion of the investigator for surgery or neoadjuvant chemotherapy. The preferred chemotherapy protocol will be FEC 100 -Taxotere (5fluorouracil 500mg/m2, Epirubicin 100 mg/m2, cyclophosphamide 500 mg/m2 (FEC) q3 weeks for 3 cycles followed by Docetaxel 100 mg/m2 (T) q 3 weeks for 3 cycles) for a total of 6 cycles with clinical and radiological assessment after each 3 cycles of chemotherapy (CT). Chemotherapy candidates will as well undergo surgery. The expected interval between the cycles will be 21 days, unless the patient has not recovered from toxicity. Specific dose adjustments will be set out in the protocol.

Breast and nodal surgery will be performed at completion of therapy (8 months of hormonal therapy for responding patients and 6 additional cycles of CT for non-responders). The type of surgery will be left at the discretion of the investigators.

Radiation therapy and adjuvant systemic treatment and endocrine therapy will be as well left at the discretion of the investigators.

Patients will be followed every 6 months during 5 years post surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to beginning specific protocol procedures including expected cooperation of the patients for the treatment and follow-up must be obtained and documented according to the local regulatory requirements.
2. Age >18.
3. Postmenopausal women or pre-menopausal (with medical or surgical oophorectomy)
4. Performance status < 2 (according to WHO criteria).
5. Histologically confirmed non-metastatic breast cancer (Luminal A or B)

   * HR (hormone receptor ) positive (Estrogen or Progesterone)> 1%.
   * Her-2 negative (score 0 or 1 by immunochemistry), FISH (fluorescence in situ hybridization) negative if IHC (immuno-histochemistry) score 2).
6. Clinical stage II and IIIa.
7. No previous breast cancer treatment by surgery, radiotherapy, hormone therapy or chemotherapy.
8. Measurable or evaluable disease.
9. Hematology:

   * Neutrophil count ≥ 1.5 G/L.
   * Platelet count ≥ 100 G/L.
   * Leucocyte count > 3.0 G/L.
   * Hb> 9g/dl.
10. Hepatic function:

    * Total bilirubin ≤ 1.5 time the Upper Normal Limit (UNL).
    * ASAT (alanine aminotransferase aspartate transaminase ) ≤ 2.5xUNL.
    * ALAT (alanine aminotransferase) ≤ 2.5xUNL.
    * Alkaline phosphatase ≤ 2.5 time the upper normal limit (UNL).
11. Renal function:

    * Serum creatinine ≤1.5xUNL (and if Serum creatinine >1.5xUNL, creatinine clearance ≥50 mL/min).
    * Creatinine clearance ≥40 mL/min in case of MRI.
12. Metabolic function:

    * Serum magnesium ≥ lower limit of normal.
    * Serum calcium ≥ lower limit of normal.
13. No progressive heart disease and no anthracycline contraindication (normal LVEF ( left ventricular ejection fraction) according to the institution guidelines).
14. Negative pregnancy test (urine or serum) within 7 days prior to registration for all women of childbearing potential. Patients of childbearing potential must implement adequate non-hormonal contraceptive measures during study treatment.

Exclusion Criteria:

1. Male patients.
2. Her-2 positive tumors or unknown HR/Her-2 status.
3. Pregnancy or breast-feeding, or plan to become pregnant within 6 months post treatment.
4. No willingness to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months post treatment.
5. Any form of breast cancer other than those described in the inclusion criteria, particularly inflammatory and/or overlooked forms (stages IIIb or IV).
6. Non-measurable tumour.
7. Bilateral breast cancer.
8. Previous treatment for breast cancer including surgery for their disease or have had primary axillary dissection, radiotherapy and systemic therapy.
9. Patient with history of other cancer, except in situ cervical cancer or baso-cellular skin cancer, considered cured.
10. Patient has another disease, which is deemed incompatible with the inclusion in the protocol.
11. Heart, kidney, medullary, respiratory or liver failure. Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 1 year before enrollment in the study.

    * History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease at baseline
    * Acute urinary infection, ongoing hemorrhagic cystitis.
12. Uncontrolled diabetes.
13. Symptomatic or progressive disorder of the central nervous system (CNS) Peripheral neuropathy > grade 2
14. Significant psychiatric abnormalities.
15. History of hypersensitivity to studied treatment or excipients
16. Known previous or ongoing abuse narcotic drug, other medication or alcohol
17. Any investigational agent within 30 days before initiation of study treatment.
18. No major surgical procedure within 28 days of initiation of treatment.
19. Subject unwilling or unable to comply with study requirement.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
pCR according to Le Chevalier's classification | up to 5 years after the end of treatment period
  pathological complete response will be assessed according to Le Chevalier's classification between two arms

SECONDARY OUTCOMES:
pCR according to Sataloff's classification | up to 5 years after the end of treatment period
  pathological complete response will be assessed according to Sataloff's classification between two arms
radiological response | up to 5 years after the end of treatment period
  radiological response according to the WHO criteria (US/Mammography/MRI)
Rate of breast conservative surgery | up to 5 years after the end of treatment period
  Rate of breast conservative surgery will be assessed and compared between two arms
Safety /Tolerability of the combination Fulvestrant + Palbociclib | up to 5 years after the end of treatment period
  Safety and tolerability will be assessed in terms of adverse events (AEs), laboratory data and vital signs. Treatment-related adverse events will be assessed by using CTCAE v4.1 classification
DFS and OS | up to 5 years after the end of treatment period
  Evaluation and comparison of Disease Free Survival (DFS) and Overall Survival (OS) between two arms

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Nabholtz, MD, Study Chair — International Cancer Research Group
Locations (14):
- Algeria (3):
  - Center Pierre et Marie Curie, Algiers
  - Cancer Center - Blida, Blida
  - CHU - Oran, Oran
- Egypt (2):
  - University of Alexandria, Alexandria
  - National Cancer Institut (NCI), Cairo
- King Hussein Cancer Center (KHCC) - Amman, Amman, Jordan
- Hotel Dieu de France, Beirut, Lebanon
- Morocco (2):
  - Hopital Cheikh Khalifa Ibn Zaid, Casablanca
  - Department of Oncology - Institut National d'Oncologie, Rabat
- Saudi Arabia (3):
  - King Abdul Aziz Medical City-National Guard Health Affairs (NGHA), Riyadh
  - Oncology Center- King Fahad Medical City (KFMC), Riyadh
  - Oncology Center- King Saud University Medical City (KSUMC), Riyadh
- Oncologie Medicale de l'Ariana (SOMA), Tunis, Tunisia
- Tawam Hospital, Al Ain City, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Alsaleh K, Al Zahwahry H, Bounedjar A, Oukkal M, Saadeddine A, Mahfouf H, Bouzid K, Bensalem A, Filali T, Abdel-Razeq H, Larbaoui B, Kandil A, Abulkhair O, Al Foheidi M, Ghosn M, Rasool H, Boussen H, Mezlini A, Haddaoui A, Ayari J, Al Ghamdi M, Errihani H, Abdel-Aziz N, Arafah M, Dabouz F, Bahadoor M, Kullab S, Nabholtz JM; King Saud University, Riyadh, Kingdom of Saudi Arabia, and the International Cancer Research Group (ICRG), Sharjah, Unites Arab Emirates. Neoadjuvant endocrine therapy with or without palbociclib in low-risk patients: a phase III randomized double-blind SAFIA trial. J Cancer Res Clin Oncol. 2023 Aug;149(9):6171-6179. doi: 10.1007/s00432-023-04588-3. Epub 2023 Jan 21. PMID 36680581